CLINICAL TRIAL: NCT05455190
Title: Parks & Pediatrics Fit Together: Translating Knowledge Into Action for Child Obesity Treatment in Partnership With Parks and Recreation
Brief Title: Parks & Pediatrics Fit Together
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00106453; 1R01HD100417-01A1 (NIH)
Record Dates: First submitted 2022-07-01; First posted 2022-07-13 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Pediatric Obesity; Implementation
Keywords: Physical Activity; Pediatrics
MeSH Terms: conditions — Pediatric Obesity; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fit Together (Experimental): Participants in the intervention arm will receive standard of care obesity treatment from their provider and be able to participate in the Fit Together program and attend activity sessions throughout the duration of their 12 month participation.
  Interventions: Behavioral: Fit Together
- Control (Active Comparator): Participants in the control arm will receive standard of care obesity treatment from their provider and a healthy cooking magazine mailed to them at a regular interval throughout the duration of their 12 month participation
  Interventions: Behavioral: Educational materials
- Fit Together - BCF Cohort (Experimental): Participants in the Fit Together - BCF Cohort arm will receive standard of care obesity treatment at the Duke Healthy Lifestyles clinic and attend Bull City Fit throughout the duration of their 6 month participation
  Interventions: Behavioral: Fit Together

INTERVENTIONS:
Behavioral: Fit Together — Fit Together intervention follows a clinic and community partnership model for childhood obesity treatment. Children with obesity will receive standard of care obesity treatment from their usual provider and will also receive a referral to an activity program run out of the local community center. Each session delivers a combination of high-intensity individual exercises, sports and games, and unstructured playtime to help children reach the US Physical Activity guidelines of 60min moderate-to-vigorous physical activity daily. There will also be a nutrition activity session offered regularly.
  Arms: Fit Together; Fit Together - BCF Cohort
Behavioral: Educational materials — Participants will receive a child-friendly cooking magazine mailed quarterly and a local Parks and Recreation program guide.
  Arms: Control

SUMMARY:
The proposed project will test an implementation strategy (the "TrailGuide") for delivering an existing model of pediatric obesity treatment ("Fit Together") that has demonstrated ability to meet published recommendations for improving health outcomes of children with obesity.

DETAILED DESCRIPTION:
Evidence-based treatment for childhood obesity exists, yet a fundamental knowledge-to-action gap has significantly limited the uptake of recommendations into clinical practice, particularly in low-income settings. Persistence of this gap represents a large-scale public health threat, as the earliest generation of children living through the obesity epidemic now enters adulthood, they are the first in US history to have a shorter life expectancy than their parents, mainly due to rising rates of obesity-related cancers and cardiovascular disease. A central challenge in delivering recommended treatment is the intensity; ≥26 hours of face-to-face contact are necessary to achieve health benefits and risk reduction. The objective of the proposed project is to develop and test an implementation strategy that pairs primary care pediatric clinics with the municipal Parks and Recreation (P&R) centers to deliver the current treatment recommendations with high fidelity, while allowing while allowing crucial adaptations for the local and cultural context. Using the Fit Together model, the clinical partner provides standard medical treatment for pediatric obesity, while the community partner (typically parks and recreation) provides space facilitating the activity/nutrition sessions specifically for children referred from the clinic, along with their families. Fit Together will be implemented in two new communities in North Carolina, and we will study implementation outcomes as well as 12-month patient outcomes. We have added a local cohort in Durham, North Carolina, where their local Fit Together model has re-started their community activity program, and we will look at 6-month patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Child receives primary care at one of the participating clinics or attends Bull City Fit
* Child age 5-12 years old at the time of enrollment in the study
* BMI greater than or equal to 95th percentile for age and sex (or greater than or equal to 85th%iile at the discretion of the provider)
* English- or Spanish-speaking

Exclusion Criteria:

* Injuries or disabilities preventing physical activity.

Inclusion criteria for caregivers:

* Age 18 or older
* English or Spanish-speaking
* Caregiver has smartphone and is willing to download app(s) used in the study
* Anticipates bringing the child to the program the majority of the time and spends significant time with the child outside of program hours (necessary in order to accurately answer survey questions about child behavior and child participation in the program, and provide feedback about the program)
* Does not have plans to leave the area during the duration of the study (12 months for Winston Salem/Charlotte participants, 6 months for Bull City Fit cohort)

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in percent of the 95th percentile for BMI Collected from clinic records. | Baseline, 6 months, and 12 months
  Change in child's BMI, based on percent of the 95th percentile, measured using height and weight collected from clinic/medical records
Proportion of children with 26 hours or more of intervention contact | Up to 12 months
  Measured by program attendance
Change in number of combined minutes per day of moderate and vigorous physical activity, as measured by Garmin vivofit4 fitness tracker | Baseline up to 12 months
  Change in physical activity measured by Garmin vivofit4 fitness tracker

SECONDARY OUTCOMES:
Change in self-report physical activity | Baseline, 6 months, and 12 months
  Measured by the Evaluation of Activity Surveys in Youth (EASY); Scoring: range 0-88, higher scores indicate more activity
Change in quality of life | Baseline, 6 months, and 12 months
  Measured by Sizing Them Up; Scoring: range 0-100, higher scores indicate better health-related quality of life
Unintended Consequences as measured by adverse events | Up to 12 months
  Measured by collecting adverse events throughout participation
Patient Satisfaction at 6 months | 6 months
  Measured by satisfaction survey; Scoring: ranging 5-25, higher scores indicate higher satisfaction
Patient Satisfaction at 12 months | 12 months
  Measured by satisfaction survey; Scoring: ranging 5-25, higher scores indicate higher satisfaction
Change in diet quality | Baseline, 6 months, 12 months
  Measured by the Dietary Screener Questionnaire (DSQ)
Healthcare utilization | Up to 12 months
  Measured by electronic health records
Cost effects | Throughout program implementation duration (approx. 30 months)
  Cost impact (summative or incremental) to the unit or organization resulting from changes in health care utilization and efficiency. Fixed and variable costs; offsets of the cost of implementation. Collected as project administrative data, surveys with clinics and P&R sites to assess additional costs.

OTHER OUTCOMES:
Fidelity | Throughout program implementation duration (approx. 30 months)
  Degree to which the program was implemented as intended. Collected via structured observations of program sessions using System for Observing Play and Leisure Activity in Youth (SOPLAY)
Implementation characteristics | Throughout program implementation duration (approx. 30 months)
  Barriers and facilitators to implementation collected via survey and qualitative interviews with stakeholders
Assessment of harms related to the program | Up through 12 months
  Measured by assessment of harms survey; Scoring: ranging 5-25, higher scores indicate higher harms
Change in mental health | Baseline, 6 months, 12 months
  Measured by Pediatric Symptom Checklist (PSC-17); Scoring: range 0-34, higher scores can indicate increased likelihood of behavioral health disorder
Change in blood pressure | Baseline, 6 months, 12 months
  Obtained from medical records
Proportion of eligible children referred to the intervention | Up through end of enrollment period (approx. 18 months)
  Proportion of eligible children who are referred to the intervention, collected via program tracking materials/referrals received and EHR

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Michael Jordan Family Medical Clinic (Freedom Drive Location) (NHPMCF), Charlotte, North Carolina
  - Waughtown Pediatrics (NHFMCF), Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] D'Agostino EM, Rosenberg LM, Richmond A, Damman A, Brown-Lowery C, Abbot-Grimes P, Siddiqui S, Fadika T, Ward M, Cooper M, Sutton S, Kenton L, Spaziano B, Kasper J, Barnes N, Hornik C. You & Me: Test and Treat study protocol for promoting COVID-19 test and treatment access to underserved populations. BMC Public Health. 2023 Oct 28;23(1):2121. doi: 10.1186/s12889-023-16960-6. PMID 37898741
- [Derived] Neshteruk CD, Skinner AC, Counts J, D'Agostino EM, Frerichs L, Howard J, Story M, Armstrong SC. Translating knowledge into action for child obesity treatment in partnership with Parks and Recreation: study protocol for a hybrid type II trial. Implement Sci. 2023 Feb 24;18(1):6. doi: 10.1186/s13012-023-01264-5. PMID 36829237